CLINICAL TRIAL: NCT04844151
Title: Acute Myocarditis Registry With Prognostic, Histologic, Immunologic, Biological, Imaging and Clinical Assessment
Acronym: AMPHIBIA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201197
Record Dates: First submitted 2021-02-24; First posted 2021-04-14 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Myocarditis
Keywords: Cardiomyopathies; Inflammatory heart disease; Magnetic resonance imaging; Viral
MeSH Terms: conditions — Myocarditis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Whole blood 20ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute myocarditis: Patients hospitalized for an acute myocarditis.

SUMMARY:
The AMPHIBIA study is an observational ambispective and prospective cohort that aim to describe the histologic, immunologic, biological, imaging, genetic and clinical characteristics of the patients hospitalized for an acute myocarditis and to evaluate their association with prognosis.

DETAILED DESCRIPTION:
Acute myocarditis is an inflammatory disease of the heart muscle. Its clinical presentation and its etiologies are multiple and make it a complex disease to treat. Its course also varies, ranging from complete clinical recovery to recurrence of ventricular arrhythmia or progression to chronic dilated heart disease, while being difficult to predict. The long-term prognosis is poorly understood.

Consecutive patients hospitalized in a tertiary university referral center cohort from 2006 to 2041 for an acute myocarditis will be ambispectively or prospectively analyzed. This project will establish a registry including up to 400 patients in the ambispective analysis cohort from 2006 to 2021 and 1000 patients in the prospective analysis cohort during a 20 years inclusion period.

The aim of the study is to describe the characteristics of patients hospitalized for an acute myocarditis and to evaluate their association wih the long term (until 20 years) prognosis.

Features of interest will include :

* Clinical
* Biological
* Etiological
* Echocardiographic
* Cardiac magnetic resonance imaging
* Genetics (for the prospective cohort)
* Anatomopathological

The collection of clinical, biological and radiological data will represent an unique source allowing research teams in the coming years to access the data necessary to answer various specific questions (pathophysiological, diagnostic, prognostic) relevant to the state of knowledge on this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocarditis confirmed by cardiac magnetic resonance according to Lake Louise modified criteria or by endomyocardial biopsy according to histologic, immunologic and immunohistochemic criteria.
* affiliation to the French Health Care System "Sécurité sociale"

Exclusion Criteria:

* Severe valvulopathy
* Complex congenital cardiopathy
* Previous heart transplant
* Known significative coronary disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalised at Pitié-Salpêtrière hospital (Paris, France) for an acute myocarditis.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2041-05-01 (Estimated); Study Completion 2041-05-01 (Estimated)

PRIMARY OUTCOMES:
Major cardiac events | up to 1 years
  Defined as a composite of :
  * All cause death
  * Resuscitated cardiac arrest
  * Heart transplant
  * Longterm mechanical circulatory support
  * Ventricular arrhythmia after discharge
  * Hospitalization for heart failure
  * Hospitalization for myocarditis recurrence

SECONDARY OUTCOMES:
Major cardiac events | up to 20 years
  Defined as a composite of :
  * All cause death
  * Resuscitated cardiac arrest
  * Heart transplant
  * Longterm mechanical circulatory support
  * Ventricular arrhythmia after discharge
  * Hospitalization for heart failure
  * Hospitalization for myocarditis recurrence
All cause death | up to 20 years
Cardiovascular death | up to 20 years
Heart transplant | up to 20 years
  Number of patients with heart transplant
Sustained ventricular arrhythmia after discharge | up to 20 years
  Number of patients with sustained ventricular arrhythmia after discharge
Resuscitated cardiac arrest | up to 20 years
  Number of patients with resuscitated cardiac arrest
Longterm mechanical circulatory support | up to 20 years
  Number of patients implanted with a longterm mechanical circulatory support
Hospitalization for myocarditis recurrence | up to 20 years
  Number of patients hospitalized for myocarditis recurrence
Hospitalization for heart failure | up to 20 years
  Number of patients with hospitalization for heart failure
Pericardial drainage | up to 20 years
  Number of patients with a surgery of pericardial drainage
Supra ventricular arrythmia | up to 20 years
  Number of patients with a new onset of supra ventricular arrhythmia
High grade atrioventricular block | up to 20 years
  Number of patients with a new high grade atrioventricular block
Pericarditis | up to 20 years
  Number of patients with pericarditis diagnosed by the patient referring physician's
Left ventricular systolic function under 50% | up to 20 years
  Evaluated by transthoracic echocardiography
Therapeutics during hospital stay | From the day of admission up to 90 days
  Type and duration of therapeutics received during the initial hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Giles MONTALESCOT, MD, PhD, Study Director — ACTION Study Group - Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Corrado D, Basso C, Thiene G. Sudden cardiac death in young people with apparently normal heart. Cardiovasc Res. 2001 May;50(2):399-408. doi: 10.1016/s0008-6363(01)00254-1. PMID 11334844
- [Background] Harmon KG, Drezner JA, Maleszewski JJ, Lopez-Anderson M, Owens D, Prutkin JM, Asif IM, Klossner D, Ackerman MJ. Pathogeneses of sudden cardiac death in national collegiate athletic association athletes. Circ Arrhythm Electrophysiol. 2014 Apr;7(2):198-204. doi: 10.1161/CIRCEP.113.001376. Epub 2014 Mar 1. PMID 24585715
- [Background] Towbin JA, Lowe AM, Colan SD, Sleeper LA, Orav EJ, Clunie S, Messere J, Cox GF, Lurie PR, Hsu D, Canter C, Wilkinson JD, Lipshultz SE. Incidence, causes, and outcomes of dilated cardiomyopathy in children. JAMA. 2006 Oct 18;296(15):1867-76. doi: 10.1001/jama.296.15.1867. PMID 17047217
- [Background] Bock CT, Klingel K, Kandolf R. Human parvovirus B19-associated myocarditis. N Engl J Med. 2010 Apr 1;362(13):1248-9. doi: 10.1056/NEJMc0911362. No abstract available. PMID 20357294
- [Background] Kuhl U, Pauschinger M, Noutsias M, Seeberg B, Bock T, Lassner D, Poller W, Kandolf R, Schultheiss HP. High prevalence of viral genomes and multiple viral infections in the myocardium of adults with "idiopathic" left ventricular dysfunction. Circulation. 2005 Feb 22;111(7):887-93. doi: 10.1161/01.CIR.0000155616.07901.35. Epub 2005 Feb 7. PMID 15699250
- [Background] Klingel K, Hohenadl C, Canu A, Albrecht M, Seemann M, Mall G, Kandolf R. Ongoing enterovirus-induced myocarditis is associated with persistent heart muscle infection: quantitative analysis of virus replication, tissue damage, and inflammation. Proc Natl Acad Sci U S A. 1992 Jan 1;89(1):314-8. doi: 10.1073/pnas.89.1.314. PMID 1309611
- [Background] Chow LH, Beisel KW, McManus BM. Enteroviral infection of mice with severe combined immunodeficiency. Evidence for direct viral pathogenesis of myocardial injury. Lab Invest. 1992 Jan;66(1):24-31. PMID 1309927
- [Background] Caforio AL, Calabrese F, Angelini A, Tona F, Vinci A, Bottaro S, Ramondo A, Carturan E, Iliceto S, Thiene G, Daliento L. A prospective study of biopsy-proven myocarditis: prognostic relevance of clinical and aetiopathogenetic features at diagnosis. Eur Heart J. 2007 Jun;28(11):1326-33. doi: 10.1093/eurheartj/ehm076. Epub 2007 May 9. PMID 17493945
- [Background] Leone O, Veinot JP, Angelini A, Baandrup UT, Basso C, Berry G, Bruneval P, Burke M, Butany J, Calabrese F, d'Amati G, Edwards WD, Fallon JT, Fishbein MC, Gallagher PJ, Halushka MK, McManus B, Pucci A, Rodriguez ER, Saffitz JE, Sheppard MN, Steenbergen C, Stone JR, Tan C, Thiene G, van der Wal AC, Winters GL. 2011 consensus statement on endomyocardial biopsy from the Association for European Cardiovascular Pathology and the Society for Cardiovascular Pathology. Cardiovasc Pathol. 2012 Jul-Aug;21(4):245-74. doi: 10.1016/j.carpath.2011.10.001. Epub 2011 Dec 3. PMID 22137237
- [Background] Aretz HT, Billingham ME, Edwards WD, Factor SM, Fallon JT, Fenoglio JJ Jr, Olsen EG, Schoen FJ. Myocarditis. A histopathologic definition and classification. Am J Cardiovasc Pathol. 1987 Jan;1(1):3-14. No abstract available. PMID 3455232
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] Anderson L, Pennell D. The role of endomyocardial biopsy in the management of cardiovascular disease: a scientific statement from the American Heart Association, the American College of Cardiology, and the European Society of Cardiology. Eur Heart J. 2008 Jul;29(13):1696; author reply 1696-7. doi: 10.1093/eurheartj/ehn189. Epub 2008 May 2. No abstract available. PMID 18456711
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Background] Ammirati E, Cipriani M, Moro C, Raineri C, Pini D, Sormani P, Mantovani R, Varrenti M, Pedrotti P, Conca C, Mafrici A, Grosu A, Briguglia D, Guglielmetto S, Perego GB, Colombo S, Caico SI, Giannattasio C, Maestroni A, Carubelli V, Metra M, Lombardi C, Campodonico J, Agostoni P, Peretto G, Scelsi L, Turco A, Di Tano G, Campana C, Belloni A, Morandi F, Mortara A, Ciro A, Senni M, Gavazzi A, Frigerio M, Oliva F, Camici PG; Registro Lombardo delle Miocarditi. Clinical Presentation and Outcome in a Contemporary Cohort of Patients With Acute Myocarditis: Multicenter Lombardy Registry. Circulation. 2018 Sep 11;138(11):1088-1099. doi: 10.1161/CIRCULATIONAHA.118.035319. PMID 29764898
- [Background] Grun S, Schumm J, Greulich S, Wagner A, Schneider S, Bruder O, Kispert EM, Hill S, Ong P, Klingel K, Kandolf R, Sechtem U, Mahrholdt H. Long-term follow-up of biopsy-proven viral myocarditis: predictors of mortality and incomplete recovery. J Am Coll Cardiol. 2012 May 1;59(18):1604-15. doi: 10.1016/j.jacc.2012.01.007. Epub 2012 Feb 22. PMID 22365425
- [Background] Aquaro GD, Perfetti M, Camastra G, Monti L, Dellegrottaglie S, Moro C, Pepe A, Todiere G, Lanzillo C, Scatteia A, Di Roma M, Pontone G, Perazzolo Marra M, Barison A, Di Bella G; Cardiac Magnetic Resonance Working Group of the Italian Society of Cardiology. Cardiac MR With Late Gadolinium Enhancement in Acute Myocarditis With Preserved Systolic Function: ITAMY Study. J Am Coll Cardiol. 2017 Oct 17;70(16):1977-1987. doi: 10.1016/j.jacc.2017.08.044. PMID 29025554
- [Background] Aquaro GD, Ghebru Habtemicael Y, Camastra G, Monti L, Dellegrottaglie S, Moro C, Lanzillo C, Scatteia A, Di Roma M, Pontone G, Perazzolo Marra M, Barison A, Di Bella G; "Cardiac Magnetic Resonance" Working Group of the Italian Society of Cardiology. Prognostic Value of Repeating Cardiac Magnetic Resonance in Patients With Acute Myocarditis. J Am Coll Cardiol. 2019 Nov 19;74(20):2439-2448. doi: 10.1016/j.jacc.2019.08.1061. PMID 31727281
- [Background] Grani C, Biere L, Eichhorn C, Kaneko K, Agarwal V, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Incremental value of extracellular volume assessment by cardiovascular magnetic resonance imaging in risk stratifying patients with suspected myocarditis. Int J Cardiovasc Imaging. 2019 Jun;35(6):1067-1078. doi: 10.1007/s10554-019-01552-6. Epub 2019 Feb 12. PMID 30756221
- [Background] Li HS, Ligons DL, Rose NR. Genetic complexity of autoimmune myocarditis. Autoimmun Rev. 2008 Jan;7(3):168-73. doi: 10.1016/j.autrev.2007.11.010. Epub 2007 Dec 3. PMID 18190873
- [Background] Rose NR, Neumann DA, Herskowitz A, Traystman MD, Beisel KW. Genetics of susceptibility to viral myocarditis in mice. Pathol Immunopathol Res. 1988;7(4):266-78. doi: 10.1159/000157122. No abstract available. PMID 2853345
- [Background] Lopez-Ayala JM, Pastor-Quirante F, Gonzalez-Carrillo J, Lopez-Cuenca D, Sanchez-Munoz JJ, Oliva-Sandoval MJ, Gimeno JR. Genetics of myocarditis in arrhythmogenic right ventricular dysplasia. Heart Rhythm. 2015 Apr;12(4):766-73. doi: 10.1016/j.hrthm.2015.01.001. Epub 2015 Jan 20. PMID 25616123